CLINICAL TRIAL: NCT03111966
Title: Effectiveness, Safety and Clinical Outcomes of Elbasvir/Grazoprevir: Results From a Spanish Real World Cohort
Status: Completed | Type: Observational
Sponsor: Hepa C (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2017-04-01; First posted 2017-04-13 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir; grazoprevir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spanish cohort with HCV treated with DAA
  Interventions: Other: Spanish cohort with HCV treated in real practice with Elbasvir/Grazoprevir

INTERVENTIONS:
Other: Spanish cohort with HCV treated in real practice with Elbasvir/Grazoprevir — Spanish cohort with HCV treated in real practice with Elbasvir/Grazoprevir

SUMMARY:
This is a multicentre, descriptive, observational and ambispective study carried out in patients who are treated with Elbasvir/Grazoprevir in hospitals that included their data in Hepa-C Registry (directed by the Spanish Association for the Study of the Liver and the Networked Biomedical Research Centre for Hepatic and Digestive Diseases).

DETAILED DESCRIPTION:
This is a multicentre, descriptive, observational and ambispective study carried out in patients who are treated with Elbasvir/Grazoprevir in hospitals that included their data in Hepa-C Registry (directed by the Spanish Association for the Study of the Liver and the Networked Biomedical Research Centre for Hepatic and Digestive Diseases)

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years to 100 years (adult).
* Sexes: all
* Healthy volunteers: no
* Chronic hepatitis C (anti-HCV antibodies and detectable HCV-RNA).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCV who are treated in real practice with Elbasvir/Grazoprevir
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
sustained virological response 12 weeks post-treatment (SVR12) | 12 weeks after the last dose of study drug
  Percentage of participants who achieve sustained virological response 12 weeks post-treatment (SVR12)
  • Measure: Hepatitis C virus ribonucleic acid (HCV-RNA) levels less than the lower limit of quantification.

SECONDARY OUTCOMES:
virologic failure | Up to 8 weeks while on treatment
  Percentage of patients with virologic failure during treatment
  • Measure: Percentage of patients with confirmed >=1 log10 IU/mL increase from nadir in HCV RNA at any time point during treatment or previous unquantifiable HCV up to 12 weeks after last dose of drug
SVR 12 and patients with mild fibrosis | Up to 12 weeks after last dose of study drug
  Percentage of patients with mild fibrosis who achieve sustained virological response 12 (SVR12) weeks post-treatment
  • Measure: percentage of patients with a baseline transient elastography < 6 kPa
low baseline viral load and SVR12 | Baseline and 12 weeks after the last dose of drug
  Percentage of participants with low baseline viral load who achieve sustained
  • Measure: HCV RNA levels less than the lower limit of quantification.

CONTACTS AND LOCATIONS:
Locations (1):
- HepaC, Madrid, Spain

REFERENCES:
- [Result] Hernandez-Conde M, Fernandez I, Perello C, Gallego A, Bonacci M, Pascasio JM, Romero-Gomez M, Llerena S, Fernandez-Rodriguez C, Castro Urda JL, Garcia Buey L, Carmona I, Morillas RM, Garcia ND, Gea F, Carrion JA, Castellote J, Moreno-Planas JM, Piqueras Alcol B, Molina E, Diago M, Montoliu S, de la Vega J, Menendez F, Sanchez Ruano JJ, Garcia-Samaniego J, Rosales-Zabal JM, Anton MD, Badia E, Souto-Rodriguez R, Salmeron FJ, Fernandez-Bermejo M, Figueruela B, Moreno-Palomares JJ, Calleja JL. Effectiveness and safety of elbasvir/grazoprevir therapy in patients with chronic HCV infection: Results from the Spanish HEPA-C real-world cohort. J Viral Hepat. 2019 Jan;26(1):55-64. doi: 10.1111/jvh.13008. Epub 2018 Oct 25. PMID 30265418